CLINICAL TRIAL: NCT00515177
Title: Mindfulness Versus Pharmacotherapy for Chronic Insomnia: A Pilot Study
Acronym: MVP#1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Hennepin County Medical Center, Minneapolis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0705M09301
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Results first posted 2013-03-29 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Insomnia; Primary Insomnia
Keywords: mindfulness; meditation; MBSR; mindfulness meditation; sleep; insomnia; chronic insomnia; primary insomnia; Minnesota
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Mindfulness-Based Stress Reduction; Eszopiclone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBSR (Experimental): A Mindfulness-Based Stress Reduction (MBSR) program that includes 8-weeks of group instruction in mindfulness meditation techniques followed by home practice and monitoring.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- PCT Sleeping Pills (Active Comparator): A pharmacotherapy control arm (PCT Sleeping Pills) consisting of a state-of-the-art prescription sedative hypnotic, eszopiclone - brand name LUNESTA(R), at a dose of one 3 milligram (mg) pill nightly for a duration of 8 weeks followed by use as needed (same dosage) for 3 months. This drug was approved by the Food and Drug Administration as a sedative for more than short term use.
  Interventions: Drug: eszopiclone

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — The intervention is a standardized program of mindfulness training led by an instructor. 8 weekly 2.5 hours sessions provide information on stress, cognition and health and training in a variety of mindfulness techniques including gentle yoga, body scan and sitting meditations. The program includes homework and home practice of mindfulness.
  Arms: MBSR
Drug: eszopiclone — One 3 mg tablet of eszopiclone nightly for 8-weeks followed by 3-months of "as needed" use
  Other Names: LUNESTA®
  Arms: PCT Sleeping Pills

SUMMARY:
Chronic insomnia is a major public health problem that affects about 10% of adults and is associated with serious and distressful health consequences such as depression, anxiety and reduced quality of life. Sleep medications are effective, but side effects, costs and uncertain long term efficacy call for non-pharmacologic alternatives. Mindfulness-Based Stress Reduction (MBSR), a standardized program of training in mindfulness meditation and yoga, is a promising new approach for treating chronic insomnia. MBSR was developed to facilitate adaptation to the stressors of medical illness. It is hypothesized that mindfulness training reduces arousal and unhelpful cognitions that promote and sustain chronic insomnia. The Mindfulness Versus Pharmacotherapy trial (MVP#1) is a pilot study designed to establish the feasibility and determine the optimal design for a full-scale trial comparing MBSR to prescribed sleep medication for treatment of chronic insomnia. For this pilot, we will randomize persons with primary chronic insomnia (actual sample of 30 persons) to 2 groups : 1) MBSR (8-weeks of group instruction followed by 3-months of home practice); and 2) PCT (3 mg of LUNESTA(eszopiclone) nightly for 8-weeks followed by 3-months of "as needed" use). Both groups will have telephone monitoring for side effects, adherence tracking, and objective sleep assessment by actigraphy. The primary outcomes are sleep quality, sleep quantity and insomnia severity assessed by well-validated self-report scales, objective sleep parameters measured by wrist actigraphy, depression and anxiety symptoms, health-related quality of life and workplace productivity. We hypothesize that those in the MBSR group will have improved sleep outcomes. Outcomes will be assessed at 8-weeks (the end of the active intervention phase) and 5 months follow-up. Outcomes will be compared to baseline values and measures reflecting proposed mechanisms of action to determine if clinically important impacts are likely to be obtainable in a full-scale trial. After follow-up data have been collected, participants will be invited to participate in focus groups to share their impressions of the study interventions to identify issues that could be addressed in a full-scale trial. Our long-range goal is to provide evidence-based recommendations for safe, practical and cost-effective non-pharmacologic treatment options for chronic insomnia.

DETAILED DESCRIPTION:
The NIH's 2003 National Sleep Disorders Research Plan defines insomnia as "difficulty falling asleep, difficulty staying asleep or short sleep duration, despite adequate opportunity for sleep," and estimates that it affects 30% to 40% of adults. The prevalence of chronic insomnia, defined as sleep disturbances for 4 weeks or more, sleep disruption with daytime impairment, or regular, nightly sleep difficulty, is about 10% of the general population, with higher rates among women, older adults and clinical populations. Total direct and indirect costs of insomnia are estimated to be roughly $113 billion annually. While only about 3 million of the 70 million Americans with insomnia take prescription medications, annual prescription drug costs for insomnia exceed $2.1 billion dollars.

Mindfulness-Based Stress Reduction (MBSR), a standardized group program of training in mindfulness meditation and yoga, is a promising intervention for lifelong self-management of chronic insomnia. Mindfulness meditation training has been found to improve sleep outcomes in patients with chronic illnesses. Meditation may be defined as self-regulation of attention, and mindfulness has been described as paying attention in a particular, intentional way, moment-by-moment, without judging. MBSR originated with the Stress Reduction Clinic at the University of Massachusetts Medical Center and is currently used in over 250 clinics, hospitals, and health maintenance organizations in the US and abroad (www.umassmed.edu/cfm/srp/).

MVP#1 is a pilot study to establish feasibility, refine procedures and determine the optimal design for a planned full-scale trial. An active control drug, eszopiclone which is a widely used and FDA approved prescription sleep medication, is included in the pilot to provide a benchmark for efficacy. Outcomes will evaluated to determine if clinically important impacts are likely to be obtainable in the future full-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Chronic insomnia defined as a) sleep onset latency and/or wake after sleep onset longer than 30 minutes per night, at least 3 nights per week; and b) Insomnia duration of at least 6 months, by self-report; and c) minimum of 1 daytime complaint by self-report (e.g. fatigue, mood disturbance);
* Between 18 and 65 years of age;
* English-speaking;
* Literate;
* Mentally intact;
* Interested in either medication or mind-body interventions;
* Able to attend weekly classes in a Minnesota Metro area;
* Able to comply with study sleep monitoring requirements;
* Willing to complete the informed consent process.

Exclusion Criteria:

* Sleep apnea or other primary sleep disorder suspected of being responsible for insomnia;
* Mental disorder or substance (including medications) suspected of being responsible for insomnia;
* General medical condition suspected of being responsible for the insomnia;
* Medically unstable (a hospital admission for non-elective purposes in the last 3 months or major surgery planned in the next 3 months);
* Serious preexisting mental health issues: suicidality or thought disorder/psychosis; or delirium or substance abuse;
* Treatment for depression or anxiety with initiation of therapy or dosage change within the last 6 months;
* Use of non-prescription sleep aids and unwilling or unable to discontinue these during the study;
* Use of prescription sleep medications or other medications known to affect sleep or be contraindicated with use of hypnotics, and unwilling or unable to discontinue these during the study;
* Known allergy to eszopiclone;
* Shift worker;
* Pregnant , breast-feeding or planning pregnancy in next 6 months;
* Previous cognitive behavioral therapy for insomnia or current psychotherapy;
* Prior MBSR class or regularly practicing mindfulness meditation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia R Gross, PhD, Principal Investigator — University of Minnesota; Mary Jo Kreitzer, RN, PhD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Minnesota Regional Sleep Disorders Center at Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- [Result] Gross CR, Kreitzer MJ, Reilly-Spong M, Wall M, Winbush NY, Patterson R, Mahowald M, Cramer-Bornemann M. Mindfulness-based stress reduction versus pharmacotherapy for chronic primary insomnia: a randomized controlled clinical trial. Explore (NY). 2011 Mar-Apr;7(2):76-87. doi: 10.1016/j.explore.2010.12.003. PMID 21397868

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through newspaper, radio advertisements and Internet.
Groups:
- MBSR: A Mindfulness-Based Stress Reduction (MBSR) program that includes 8-weeks of group instruction in mindfulness meditation techniques followed by home practice and monitoring.
  Mindfulness-Based Stress Reduction : The intervention is a standardized program of mindfulness training led by an instructor. 8 weekly 2.5 hours sessions provide information on stress, cognition and health and training in a variety of mindfulness techniques including gentle yoga, body scan and sitting meditations. The program includes homework and home practice of mindfulness.
- Pharmacotherapy Control Arm: A pharmacotherapy control arm (PCT) consisting of a state-of-the-art prescription sedative hypnotic, approved by the Food and Drug Administration for more than short term use.
  eszopiclone : One 3 mg tablet of eszopiclone nightly for 8-weeks followed by 3-months of "as needed" use
Period: Overall Study
Arm/Group | MBSR | Pharmacotherapy Control Arm
Started | 20 | 10
Completed | 18 | 9
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized to MBSR | Randomized to PCT | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 10 | 29
  >=65 years | 1 | 0 | 1
Age Continuous [Median (Full Range); unit: years] | 47 [21 to 65] | 53.5 [29 to 59] | 51 [21 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI is a 19-item self-reported sleep quality measure with scores that range from 0 to 21, where higher scores indicate worse sleep quality. Scores greater than 5 indicate poor sleep.
Time Frame: 8 weeks and 5 months
Population: In the PCT arm, one person who refused to take the drug was excluded. 10-1=9 In the MBSR arm, one person who did not attend MBSR and one person who attended fewer than 5 classes were excluded. 20-2=18.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBSR | Pharmacotherapy Control Arm
Number analyzed (Participants) | 18 | 9
units on a scale
  8 weeks | 7.7 (3.6) | 9.2 (2.0)
  5 months | 7.0 (4.6) | 8.2 (2.7)

2. Primary Outcome: Insomnia Severity Index
Description: The Insomnia Severity Index is a 7-item scale that provides a total score indicating current (e.g., last 2 weeks) severity of insomnia symptoms with scores that can range from 0 to 28. Scores of 15 or higher indicate clinical insomnia.
Time Frame: 8 weeks and 5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBSR | Pharmacotherapy Control Arm
Number analyzed (Participants) | 18 | 9
units on a scale
  8 week | 9.6 (4.2) | 9.1 (4.6)
  5 months | 8.1 (5.5) | 7.8 (4.3)

3. Primary Outcome: Actigraphy
Description: Total Sleep Time from Actigraphy
Time Frame: 8 weeks
Population: In the PCT arm, one person who refused to take the drug and one who did not complete actigraphy were excluded. 10-2=8 In the MBSR arm, one person who did not attend MBSR, one person who attended fewer than 5 classes, and two who did not complete actigraphy were excluded. 20-4=16.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | MBSR | Pharmacotherapy Control Arm
Number analyzed (Participants) | 16 | 8
hours | 6.2 (0.8) | 6.9 (0.6)

4. Secondary Outcome: State-Trait Anxiety Inventory (STAI)
Description: The STAI is a 20 item scale that measures current anxiety symptoms with scores that range from 20 to 80, with higher scores indicating greater levels of anxiety. The norm for working adults is a score of 34.
Time Frame: 8 weeks and 5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBSR | Pharmacotherapy Control Arm
Number analyzed (Participants) | 18 | 9
units on a scale
  8 week | 32.9 (12.0) | 31.3 (14.9)
  5 months | 30.1 (11.8) | 28.3 (8.5)

5. Secondary Outcome: Center for Epidemiological Studies Depression Scale (CES-D)
Description: The CES-D is a 20-item self-report scale to measure symptoms of depression in the past week with scores having a range of 0 to 60 and a score of 16 or higher indicating clinically relevant symptoms.
Time Frame: 8 weeks and 5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBSR | Pharmacotherapy Control Arm
Number analyzed (Participants) | 18 | 9
units on a scale
  8 week | 10.0 (8.5) | 10.1 (12.1)
  5 months | 8.4 (7.6) | 7.0 (5.8)

6. Secondary Outcome: Medical Outcome Study Short Form (SF-12)
Description: Mental component summary score (MCS) of the SF-12 is a self-reported measure of mental health-related quality of life. Scores are reported as standardized T-scores, where an average (mean) score in the general population is 50 with a standard deviation of 10. Scores of 40 or less indicate impaired mental health quality or function.
Time Frame: 8 weeks and 5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBSR | Pharmacotherapy Control Arm
Number analyzed (Participants) | 18 | 9
units on a scale
  8 week | 48.8 (8.5) | 48.3 (12.7)
  5 months | 49.7 (10.1) | 50.1 (6.7)

ADVERSE EVENTS:
Time Frame: Adverse events were queried weekly from intervention start to 12 weeks, bi-monthly in month 4, monthly in months 5 (intervention end) and 6 (post-intervention).
Description: Participants in the PCT (pharmacotherapy) arm received scheduled phone calls and were asked if they had experienced common known side-effects of their medication (e.g. headache, nausea/vomiting, excessive sleepiness, taste disturbance) or health problem since the last call.
  MBSR participants were also called weekly & asked how there health was.
Groups:
- Pharmacotherapy (Eszopiclone, 3mg): The PCT control treatment consisted of 3mg eszopiclone nightly for 8 weeks, followed by use as needed for 3 months.
- MBSR: Mindfulness-Based Stress Reduction (MBSR) is an 8 week program of yoga and mindfulness training taught by a trained instructor in a group format.
Arm/Group | Pharmacotherapy (Eszopiclone, 3mg) | MBSR
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/20
Other Adverse Events (participants affected / at risk) | 7/10 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pharmacotherapy (Eszopiclone, 3mg) (N=10) | MBSR (N=20)
Excessive sleepiness (Nervous system disorders) | 3 (9) | 0 (0)
Headache (General disorders) | 2 (7) | 0 (0)
Taste disturbance (General disorders) | 4 (12) | 0 (0) — Bitter taste
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Reflux (Gastrointestinal disorders) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Hypertension (Renal and urinary disorders) | 1 (1) | 0 (0)
Strange dreams (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes